CLINICAL TRIAL: NCT04436107
Title: A Phase 1, Open Label, Multiple Dose, Dose Escalation and Expansion Study of Bruton Tyrosine Kinase (BTK) Inhibitor, Zanubrutinib, in Combination With Lenalidomide, With or Without Rituximab in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Zanubrutinib, in Combination With Lenalidomide, With or Without Rituximab in Participants With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-110
Record Dates: First submitted 2020-06-16; First posted 2020-06-17 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Relapsed/Refractory Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1: Zanubrutinib + Lenalidomide 15 mg (Experimental): Participants received zanubrutinib 160 mg orally twice a day (BID) and lenalidomide 15 mg orally once a day (QD) on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Zanubrutinib; Drug: Lenalidomide
- Part 1: Zanubrutinib + Lenalidomide 20 mg (Experimental): Participants received zanubrutinib 160 mg orally BID and lenalidomide 20 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Zanubrutinib; Drug: Lenalidomide
- Part 1: Zanubrutinib + Lenalidomide 25 mg (Experimental): Participants received zanubrutinib 160 mg orally BID and lenalidomide 25 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Zanubrutinib; Drug: Lenalidomide
- Part 2: Zanubrutinib + Lenalidomide 25 mg (Experimental): Participants received zanubrutinib 160 mg orally BID and lenalidomide 25 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Zanubrutinib; Drug: Lenalidomide

INTERVENTIONS:
Drug: Zanubrutinib — 160 mg administered orally twice daily (BID)
  Other Names: BGB-3111; BRUKINSA
Drug: Lenalidomide — Administered orally on Days 1-21 each cycle followed by a mandatory 7-day drug-free interval.

SUMMARY:
The primary objective of this study is to determine the maximum tolerated doses (MTD) and the recommended Phase 2 dose (RP2D), and safety, tolerability, and efficacy of zanubrutinib in combination with lenalidomide in participants with R/R DLBCL

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed DLBCL, all participants must provide sufficient archival or fresh tumor tissue samples for evaluation by immunohistochemistry (IHC) and Gene Expression Profiling (GEP).
2. Relapsed or refractory disease, defined as either: 1) progression of disease after having achieved disease remission (complete response [CR] or partial response [PR]) , or 2) stable disease (SD), or progressive disease (PD) at completion of the treatment regimen preceding entry to the study.
3. Participants who have not received high dose therapy/stem cell transplantation (HDT/SCT) must be ineligible for HDT/SCT.
4. Measurable disease as defined by at least 1 lymph node >1.5 cm in longest diameter, or at least 1 extra-nodal lesion >1.0 cm in longest diameter, and measurable in 2 perpendicular dimensions.
5. Received an appropriate first-line therapy for DLBCL,defined as an anti CD20 antibody and an appropriate anthracycline-based combination therapy for at least 2 cycles, unless the patient is intolerant or had disease progression before Cycle 2..

Key Exclusion Criteria:

1. Current or history of central nervous system (CNS) lymphoma.
2. Histologically transformed lymphoma.
3. History of allogeneic stem-cell transplantation.
4. Prior exposure to a BTK inhibitor.
5. Prior exposure to lenalidomide or thalidomide.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (10):
- China (10):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Jilin Cancer Hospital, Changchun, Jilin
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 10 study centers in China. Participants with relapsed/refractory diffuse large B-cell lymphoma (R/R DLBCL) ineligible for high-dose therapy/stem cell transplant who had received ≥ 1 prior line of systemic therapy were enrolled.
Period: Overall Study
Arm/Group | Part 1: Zanubrutinib + Lenalidomide 15 mg | Part 1: Zanubrutinib + Lenalidomide 20 mg | Part 1: Zanubrutinib + Lenalidomide 25 mg | Part 2: Zanubrutinib + Lenalidomide 25 mg
Started | 6 | 10 | 11 | 39
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 10 | 11 | 39
Not completed — Sponsor Ended Study | 2 | 4 | 8 | 20
Not completed — Death | 3 | 5 | 3 | 18
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Zanubrutinib + Lenalidomide 15 mg: Participants received zanubrutinib 160 mg orally BID and lenalidomide 15 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Part 1: Zanubrutinib + Lenalidomide 15 mg | Part 1: Zanubrutinib + Lenalidomide 20 mg | Part 1: Zanubrutinib + Lenalidomide 25 mg | Part 2: Zanubrutinib + Lenalidomide 25 mg | Total
Number analyzed (Participants) | 6 | 10 | 11 | 39 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (15.12) | 54.0 (14.83) | 58.8 (13.12) | 59.1 (11.61) | 57.2 (12.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6 | 19 | 31
  Male | 4 | 6 | 5 | 20 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 10 | 11 | 39 | 66
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 6 | 10 | 11 | 39 | 66

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product (zanubrutinib in combination with lenalidomide).
  A serious adverse event (SAE) is any untoward medical occurrence that, at any dose:
  * Resulted in death.
  * Was life threatening.
  * Required hospitalization or prolongation of existing hospitalization.
  * Resulted in disability/incapacity.
  * Was a congenital anomaly/birth defect.
  * Was considered a significant medical AE by the investigator based on medical judgement (eg, may have jeopardized the patient or may have required medical/surgical intervention to prevent one of the outcomes listed above).
Time Frame: From first dose of study drug to 30 days after last dose. Maximum time on treatment in Part 1 was 1260 days.
Population: The safety analysis set was defined as all participants who received at least one dose of any medication within the combination therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Zanubrutinib + Lenalidomide 15 mg | Part 1: Zanubrutinib + Lenalidomide 20 mg | Part 1: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 6 | 10 | 11
Participants
  TEAEs | 6 | 10 | 11
  SAEs | 0 | 3 | 4

2. Primary Outcome: Part 2: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved a best overall response of partial response (PR) or complete response (CR) based on the Lugano classification as assessed by the investigator. Response was evaluated using computed tomography (CT) and metabolic imaging (fluorodeoxyglucose-positron emission tomography (FDG-PET)).
  CR: complete metabolic (no/minimal FDG uptake and no evidence of FDG-avid disease in bone marrow) and radiologic response (target lesions regressed to ≤ 1.5 cm in longest diameter with no extra-lymphatic sites of disease, no organ enlargement and normal bone marrow morphology), no new lesions, and no bone marrow involvement confirmed by bone marrow biopsies (if bone marrow was involved at baseline).
  PR is partial metabolic (reduced FDG uptake from Baseline) and radiologic response (≥ 50% decrease in size of measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by > 50% in length beyond normal) and no new lesions.
Time Frame: Response was assessed every 12 weeks for the first 48 weeks and every 16 weeks for the next 48 weeks and every 24 weeks thereafter; maximum time on follow-up was 24 months in Part 2 and 31 months in the RP2D group.
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL. Participants with no post-baseline response assessments were treated as non-responders.
  Overall response rate was a prespecified primary endpoint in Part 2 only; results are also presented for all participants (Part 1 + Part 2) who received the recommended phase 2 dose (RP2D) of lenalidomide (25 mg).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 1+2: Zanubrutinib + Lenalidomide 25 mg: All participants who received the Recommended Phase 2 dose (RP2D) of zanubrutinib 160 mg orally BID and lenalidomide 25 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
Arm/Group | Part 2: Zanubrutinib + Lenalidomide 25 mg | Part 1+2: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 39 | 50
percentage of participants | 48.7 [32.4 to 65.2] | 58.0 [43.2 to 71.8]

3. Secondary Outcome: Part 1: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved a best overall response of partial response or complete response based on the Lugano classification as assessed by the investigator. Response was evaluated using CT and metabolic imaging (FDG-PET).
  CR: complete metabolic (no/minimal FDG uptake and no evidence of FDG-avid disease in bone marrow) and radiologic response (target lesions regressed to ≤ 1.5 cm in longest diameter with no extra-lymphatic sites of disease, no organ enlargement and normal bone marrow morphology), no new lesions, and no bone marrow involvement confirmed by bone marrow biopsies (if bone marrow was involved at baseline).
  PR is partial metabolic (reduced FDG uptake from Baseline) and radiologic response (≥ 50% decrease in size of measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by > 50% in length beyond normal) and no new lesions.
Time Frame: Response was assessed every 12 weeks for the first 48 weeks and every 16 weeks for the next 48 weeks and every 24 weeks thereafter; maximum time on follow-up in Part 1 was 42 months.
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL. Participants with no post-baseline response assessments were treated as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Zanubrutinib + Lenalidomide 15 mg | Part 1: Zanubrutinib + Lenalidomide 20 mg | Part 1: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 6 | 10 | 11
percentage of participants | 16.7 [0.4 to 64.1] | 30.0 [6.7 to 65.2] | 90.9 [58.7 to 99.8]

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to 8 Hours Postdose (AUCt) of Zanubrutinib After a Single Dose and at Steady State
Description: Blood samples to characterize the pharmacokinetic (PK) profile of zanubrutinib and lenalidomide when given in combination were collected after a single dose (Cycle 1 Day 1) and at steady state (Cycle 1 Day 21) for participants in Part 1 and for twelve participants from the first stage of enrollment in Part 2.
  The lower limit of quantitation (LLOQ) was 1.00 ng/mL.
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: The PK analysis set was defined as all participants who had at least one post-dose plasma concentration collected without a major protocol deviation affecting PK. Per the prespecified analysis of zanubrutinib PK parameters, participants were analyzed in one group since there was only one dose level for zanubrutinib, regardless of dose of lenalidomide they received.
  The analysis includes participants with available PK parameter data at each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Day 1 Zanubrutinib + Lenalidomide; Day 21 Zanubrutinib + Lenalidomide: Participants received zanubrutinib 160 mg orally BID and lenalidomide orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
Arm/Group | Day 1 Zanubrutinib + Lenalidomide | Day 21 Zanubrutinib + Lenalidomide
Number analyzed (Participants) | 30 | 25
h*ng/mL | 847.8 (80) | 623.9 (49)

5. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast) of Zanubrutinib After a Single Dose and at Steady State
Description: Blood samples to characterize the PK profile of zanubrutinib and lenalidomide when given in combination were collected after first dose (Cycle 1 Day 1) and at steady state (Cycle 1 Day 21) for participants in Part 1 and for twelve participants from the first stage of enrollment in Part 2.
  The lower limit of quantitation was 1.00 ng/mL.
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Day 1 Zanubrutinib + Lenalidomide | Day 21 Zanubrutinib + Lenalidomide
Number analyzed (Participants) | 39 | 36
h*ng/mL | 798.4 (94) | 638.4 (57)

6. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf) of Zanubrutinib After a Single Dose
Description: Blood samples to characterize the PK profile of zanubrutinib and lenalidomide when given in combination were collected after first dose (Cycle 1 Day 1) for participants in Part 1 and for twelve participants from the first stage of enrollment in Part 2.
  The lower limit of quantitation was 1.00 ng/mL.
Time Frame: Cycle 1 Day 1, 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: The PK analysis set was defined as all participants who had at least one post-dose plasma concentration collected without a major protocol deviation affecting PK. Per the prespecified analysis of zanubrutinib PK parameters, participants were analyzed in one group since there was only one dose level for zanubrutinib, regardless of dose of lenalidomide they received.
  The analysis includes participants with available AUCinf data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Day 1 Zanubrutinib + Lenalidomide
Number analyzed (Participants) | 21
h*ng/mL | 943.3 (81)

7. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Zanubrutinib After a Single Dose and at Steady State
Description: as for outcome 5
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Day 1 Zanubrutinib + Lenalidomide | Day 21 Zanubrutinib + Lenalidomide
Number analyzed (Participants) | 39 | 36
ng/mL | 281.2 (85) | 208.7 (61)

8. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Zanubrutinib After a Single Dose and at Steady State
Description: as for outcome 5
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Day 1 Zanubrutinib + Lenalidomide | Day 21 Zanubrutinib + Lenalidomide
Number analyzed (Participants) | 39 | 36
hours | 2.0 [0.9 to 8.0] | 2.5 [0.4 to 8.0]

9. Secondary Outcome: Time to the Last Quantifiable Concentration (Tlast) of Zanubrutinib After a Single Dose and at Steady State
Description: as for outcome 5
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Day 1 Zanubrutinib + Lenalidomide | Day 21 Zanubrutinib + Lenalidomide
Number analyzed (Participants) | 39 | 36
hours | 7.9 [7.5 to 8.2] | 7.9 [7.5 to 8.1]

10. Secondary Outcome: Apparent Terminal Elimination Half-life (T1/2) of Zanubrutinib After a Single Dose and at Steady State
Description: as for outcome 4
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: as for outcome 4
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | Day 1 Zanubrutinib + Lenalidomide | Day 21 Zanubrutinib + Lenalidomide
Number analyzed (Participants) | 22 | 18
hours | 1.4 [0.9 to 3.1] | 1.6 [1.1 to 3.0]

11. Secondary Outcome: Apparent Volume (CL/F) of Zanubrutinib After a Single Dose and at Steady State
Description: as for outcome 4
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Day 1 Zanubrutinib + Lenalidomide | Day 21 Zanubrutinib + Lenalidomide
Number analyzed (Participants) | 22 | 18
L/h | 165.9 (80) | 226.5 (46)

12. Secondary Outcome: Apparent Clearance (Vz/F) of Zanubrutinib After a Single Dose and at Steady State
Description: as for outcome 4
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Day 1 Zanubrutinib + Lenalidomide | Day 21 Zanubrutinib + Lenalidomide
Number analyzed (Participants) | 22 | 18
liters | 341.4 (69) | 533.8 (54)

13. Secondary Outcome: Accumulation Ratio of AUCt for Zanubrutinib
Description: Blood samples to characterize the pharmacokinetic (PK) profile of zanubrutinib and lenalidomide when given in combination were collected after a single dose (Cycle 1 Day 1) and at steady state (Cycle 1 Day 21) for participants in Part 1 and for twelve participants from the first stage of enrollment in Part 2.
  The lower limit of quantitation (LLOQ) was 1.00 ng/mL. Accumulation ratio is defined as the ratio of AUCt at steady state (Day 21) to the AUCt after the first dose (Day 1).
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: The PK analysis set was defined as all participants who had at least one post-dose plasma concentration collected without a major protocol deviation affecting PK. Per the prespecified analysis of zanubrutinib PK parameters, participants were analyzed in one group since there was only one dose level for zanubrutinib, regardless of dose of lenalidomide they received. The analysis includes participants with available AUCt data at both Day 1 and Day 21.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Groups:
- Zanubrutinib + Lenalidomide: Participants received zanubrutinib 160 mg orally BID and lenalidomide orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
Arm/Group | Zanubrutinib + Lenalidomide
Number analyzed (Participants) | 23
ratio | 0.7 (50)

14. Secondary Outcome: Accumulation Ratio of Cmax for Zanubrutinib
Description: Blood samples to characterize the pharmacokinetic (PK) profile of zanubrutinib and lenalidomide when given in combination were collected after a single dose (Cycle 1 Day 1) and at steady state (Cycle 1 Day 21) for participants in Part 1 and for twelve participants from the first stage of enrollment in Part 2.
  The lower limit of quantitation (LLOQ) was 1.00 ng/mL. Accumulation ratio is defined as the ratio of Cmax at steady state (Day 21) to the Cmax after the first dose (Day 1).
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: The PK analysis set was defined as all participants who had at least one post-dose plasma concentration collected without a major protocol deviation affecting PK. Per the prespecified analysis of zanubrutinib PK parameters, participants were analyzed in one group since there was only one dose level for zanubrutinib, regardless of dose of lenalidomide they received. The analysis includes participants with available Cmax data at both Day 1 and Day 21.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Zanubrutinib + Lenalidomide
Number analyzed (Participants) | 36
ratio | 0.8 (73)

15. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to 8 Hours Postdose (AUCt) of Lenalidomide After a Single Dose and at Steady State
Description: Blood samples to characterize the pharmacokinetic (PK) profile of zanubrutinib and lenalidomide when given in combination were collected after a single dose (Cycle 1 Day 1) and at steady state (Cycle 1 Day 21) for participants in Part 1 and for twelve participants from the first stage of enrollment in Part 2.
  The lower limit of quantitation was 2.00 ng/mL.
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: The PK analysis set was defined as all participants who had at least one post-dose plasma concentration collected without a major protocol deviation affecting PK.
  The analysis includes participants with available PK parameter data at each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Day 1 Zanubrutinib + Lenalidomide 15 mg; Day 21 Zanubrutinib + Lenalidomide 15 mg: Participants received zanubrutinib 160 mg orally BID and lenalidomide 15 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- Day 1 Zanubrutinib + Lenalidomide 20 mg; Day 21 Zanubrutinib + Lenalidomide 20 mg: Participants received zanubrutinib 160 mg orally BID and lenalidomide 20 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- Day 1 Zanubrutinib + Lenalidomide 25 mg; Day 21 Zanubrutinib + Lenalidomide 25 mg: Participants received zanubrutinib 160 mg orally BID and lenalidomide 25 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
Arm/Group | Day 1 Zanubrutinib + Lenalidomide 15 mg | Day 1 Zanubrutinib + Lenalidomide 20 mg | Day 1 Zanubrutinib + Lenalidomide 25 mg | Day 21 Zanubrutinib + Lenalidomide 15 mg | Day 21 Zanubrutinib + Lenalidomide 20 mg | Day 21 Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 5 | 9 | 20 | 2 | 7 | 15
h*ng/mL | 843.5 (51) | 1092.5 (59) | 1177.7 (125) | 1091.0 (34) | 916.1 (39) | 1702.6 (29)

16. Secondary Outcome: AUClast of Lenalidomide After a Single Dose and at Steady State
Description: as for outcome 15
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Day 1 Zanubrutinib + Lenalidomide 15 mg | Day 1 Zanubrutinib + Lenalidomide 20 mg | Day 1 Zanubrutinib + Lenalidomide 25 mg | Day 21 Zanubrutinib + Lenalidomide 15 mg | Day 21 Zanubrutinib + Lenalidomide 20 mg | Day 21 Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 6 | 10 | 23 | 3 | 9 | 20
h*ng/mL | 641.9 (91) | 1072.7 (56) | 1187.4 (112) | 778.7 (69) | 824.6 (41) | 1389.7 (53)

17. Secondary Outcome: AUCinf of Lenalidomide After a Single Dose
Description: as for outcome 15
Time Frame: Cycle 1 Day 1 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Day 1 Zanubrutinib + Lenalidomide 15 mg | Day 1 Zanubrutinib + Lenalidomide 20 mg | Day 1 Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 5 | 6 | 14
h*ng/mL | 933.7 (52) | 1443.2 (29) | 1752.4 (28)

18. Secondary Outcome: Cmax of Lenalidomide After a Single Dose and at Steady State
Description: as for outcome 15
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Day 1 Zanubrutinib + Lenalidomide 15 mg | Day 1 Zanubrutinib + Lenalidomide 20 mg | Day 1 Zanubrutinib + Lenalidomide 25 mg | Day 21 Zanubrutinib + Lenalidomide 15 mg | Day 21 Zanubrutinib + Lenalidomide 20 mg | Day 21 Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 6 | 10 | 23 | 3 | 9 | 20
ng/mL | 206.4 (118) | 276.5 (68) | 332.0 (123) | 238.5 (132) | 206.6 (57) | 372.1 (67)

19. Secondary Outcome: Tmax of Lenalidomide After a Single Dose and at Steady State
Description: as for outcome 15
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | Day 1 Zanubrutinib + Lenalidomide 15 mg | Day 1 Zanubrutinib + Lenalidomide 20 mg | Day 1 Zanubrutinib + Lenalidomide 25 mg | Day 21 Zanubrutinib + Lenalidomide 15 mg | Day 21 Zanubrutinib + Lenalidomide 20 mg | Day 21 Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 6 | 10 | 23 | 3 | 9 | 20
hours | 1.5 [0.5 to 7.6] | 1.5 [0.9 to 4.3] | 2.0 [0.5 to 4.1] | 1.9 [0.5 to 3.8] | 2.1 [0.6 to 4.0] | 1.9 [0.4 to 7.9]

20. Secondary Outcome: Tlast of Lenalidomide After a Single Dose and at Steady State
Description: as for outcome 15
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | Day 1 Zanubrutinib + Lenalidomide 15 mg | Day 1 Zanubrutinib + Lenalidomide 20 mg | Day 1 Zanubrutinib + Lenalidomide 25 mg | Day 21 Zanubrutinib + Lenalidomide 15 mg | Day 21 Zanubrutinib + Lenalidomide 20 mg | Day 21 Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 6 | 10 | 23 | 3 | 9 | 20
hours | 7.6 [7.6 to 8.0] | 7.9 [7.6 to 8.2] | 8.0 [7.5 to 8.1] | 7.7 [7.5 to 7.9] | 7.7 [7.5 to 8.1] | 8.0 [7.5 to 8.1]

21. Secondary Outcome: T1/2 of Lenalidomide After a Single Dose and at Steady State
Description: as for outcome 15
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: as for outcome 15
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | Day 1 Zanubrutinib + Lenalidomide 15 mg | Day 1 Zanubrutinib + Lenalidomide 20 mg | Day 1 Zanubrutinib + Lenalidomide 25 mg | Day 21 Zanubrutinib + Lenalidomide 15 mg | Day 21 Zanubrutinib + Lenalidomide 20 mg | Day 21 Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 5 | 8 | 17 | 2 | 6 | 14
hours | 2.3 [2.0 to 2.6] | 2.7 [1.7 to 3.9] | 2.5 [1.7 to 7.7] | 2.0 [1.8 to 2.2] | 2.3 [2.0 to 2.9] | 2.4 [1.9 to 3.4]

22. Secondary Outcome: CL/F of Lenalidomide After a Single Dose and at Steady State
Description: as for outcome 15
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Day 1 Zanubrutinib + Lenalidomide 15 mg | Day 1 Zanubrutinib + Lenalidomide 20 mg | Day 1 Zanubrutinib + Lenalidomide 25 mg | Day 21 Zanubrutinib + Lenalidomide 15 mg | Day 21 Zanubrutinib + Lenalidomide 20 mg | Day 21 Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 5 | 8 | 17 | 2 | 6 | 14
L/h | 16.1 (52) | 16.0 (52) | 13.9 (41) | 12.8 (35) | 17.6 (36) | 12.5 (31)

23. Secondary Outcome: Vz/F of Lenalidomide After a Single Dose and at Steady State
Description: as for outcome 15
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Day 1 Zanubrutinib + Lenalidomide 15 mg | Day 1 Zanubrutinib + Lenalidomide 20 mg | Day 1 Zanubrutinib + Lenalidomide 25 mg | Day 21 Zanubrutinib + Lenalidomide 15 mg | Day 21 Zanubrutinib + Lenalidomide 20 mg | Day 21 Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 5 | 8 | 17 | 2 | 6 | 14
liters | 53.6 (42) | 62.1 (76) | 49.7 (49) | 37.3 (19) | 57.6 (28) | 43.6 (20)

24. Secondary Outcome: Accumulation Ratio of AUCt for Lenalidomide
Description: Blood samples to characterize the pharmacokinetic (PK) profile of zanubrutinib and lenalidomide when given in combination were collected after a single dose (Cycle 1 Day 1) and at steady state (Cycle 1 Day 21) for participants in Part 1 and for twelve participants from the first stage of enrollment in Part 2.
  The lower limit of quantitation was 2.00 ng/mL. Accumulation ratio is defined as the ratio of AUCt at steady state (Day 21) to AUCt after the first dose (Day 1).
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: The PK analysis set was defined as all participants who had at least one post-dose plasma concentration collected without a major protocol deviation affecting PK.
  The analysis includes participants with available AUCt data at both Day 1 and Day 21.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Groups:
- Zanubrutinib + Lenalidomide 15 mg: Participants received zanubrutinib 160 mg orally BID and lenalidomide 15 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- Zanubrutinib + Lenalidomide 20 mg: Participants received zanubrutinib 160 mg orally BID and lenalidomide 20 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- Zanubrutinib + Lenalidomide 25 mg: Participants received zanubrutinib 160 mg orally BID and lenalidomide 25 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
Arm/Group | Zanubrutinib + Lenalidomide 15 mg | Zanubrutinib + Lenalidomide 20 mg | Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 2 | 6 | 13
ratio | 1.1 (48) | 0.8 (106) | 1.0 (27)

25. Secondary Outcome: Accumulation Ratio of Cmax for Lenalidomide
Description: Blood samples to characterize the pharmacokinetic (PK) profile of zanubrutinib and lenalidomide when given in combination were collected after a single dose (Cycle 1 Day 1) and at steady state (Cycle 1 Day 21) for participants in Part 1 and for twelve participants from the first stage of enrollment in Part 2.
  The lower limit of quantitation was 2.00 ng/mL. Accumulation ratio is defined as the ratio of Cmax at steady state (Day 21) to Cmax after the first dose (Day 1).
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 21 at predose and 0.5, 1, 2, 3, 4, and 8 hours postdose
Population: The PK analysis set was defined as all participants who had at least one post-dose plasma concentration collected without a major protocol deviation affecting PK.
  The analysis includes participants with available Cmax data at both Day 1 and Day 21.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Zanubrutinib + Lenalidomide 15 mg | Zanubrutinib + Lenalidomide 20 mg | Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 3 | 9 | 20
ratio | 1.3 (51) | 0.8 (100) | 0.9 (59)

26. Secondary Outcome: Part 1: Overall Response Rate by Immunohistochemistry Subtypes
Description: ORR is defined as the percentage of participants who achieved a best overall response of PR or CR based on the Lugano classification as assessed by the investigator. Response was evaluated using CT and metabolic imaging (FDG-PET).
  CR: complete metabolic (no/minimal FDG uptake and no evidence of FDG-avid disease in bone marrow) and radiologic response (target lesions regressed to ≤ 1.5 cm in longest diameter with no extra-lymphatic sites of disease, no organ enlargement and normal bone marrow morphology), no new lesions, and no bone marrow involvement confirmed by bone marrow biopsies (if bone marrow was involved at baseline).
  PR is partial metabolic (reduced FDG uptake from Baseline) and radiologic response (≥ 50% decrease in size of measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by > 50% in length beyond normal) and no new lesions.
  Immunohistochemistry (IHC) was used to identify germinal B-cell-like (GCB) and non-GCB phenotypes.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- GCB Subtype: Zanubrutinib + Lenalidomide 15 mg: Participants with IHC GCB subtype received zanubrutinib 160 mg orally BID and lenalidomide 15 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- Non-GCB Subtype: Zanubrutinib + Lenalidomide 15 mg: Participants with IHC non-GCB subtype received zanubrutinib 160 mg orally BID and lenalidomide 15 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- GCB Subtype: Zanubrutinib + Lenalidomide 20 mg: Participants with IHC GCB subtype received zanubrutinib 160 mg orally BID and lenalidomide 20 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- Non-GCB Subtype: Zanubrutinib + Lenalidomide 20 mg: Participants with IHC non-GCB subtype received zanubrutinib 160 mg orally BID and lenalidomide 20 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- GCB Subtype: Zanubrutinib + Lenalidomide 25 mg: Participants in Part 1 with IHC GCB subtype received zanubrutinib 160 mg orally BID and lenalidomide 25 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- Non-GCB Subtype: Zanubrutinib + Lenalidomide 25 mg: Participants in Part 1 with IHC non-GCB subtype received zanubrutinib 160 mg orally BID and lenalidomide 25 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
Arm/Group | GCB Subtype: Zanubrutinib + Lenalidomide 15 mg | Non-GCB Subtype: Zanubrutinib + Lenalidomide 15 mg | GCB Subtype: Zanubrutinib + Lenalidomide 20 mg | Non-GCB Subtype: Zanubrutinib + Lenalidomide 20 mg | GCB Subtype: Zanubrutinib + Lenalidomide 25 mg | Non-GCB Subtype: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 3 | 3 | 4 | 6 | 3 | 8
percentage of participants | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 50.0 [6.8 to 93.2] | 16.7 [0.4 to 64.1] | 66.7 [9.4 to 99.2] | 100.0 [63.1 to 100.0]

27. Secondary Outcome: Part 1: Overall Response Rate by Gene Expression Profiling (GEP) Subtypes
Description: The percentage of participants who achieved a best overall response of PR or CR based on the Lugano classification as assessed by the investigator. Response was evaluated using CT and metabolic imaging.
  CR: complete metabolic (no/minimal FDG uptake and no evidence of FDG-avid disease in bone marrow) and radiologic response (target lesions regressed to ≤ 1.5 cm in longest diameter with no extra-lymphatic sites of disease, no organ enlargement and normal bone marrow morphology), no new lesions, and no bone marrow involvement confirmed by bone marrow biopsies (if bone marrow was involved at baseline).
  PR: partial metabolic (reduced FDG uptake from Baseline) and radiologic response (≥ 50% decrease in size of measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by > 50% in length beyond normal) and no new lesions.
  Gene expression profiling by HTG EdgeSeq DLBCL cell-of-origin (COO) assay was used to determine activated B-cell like (ABC) and GCB subtypes.
Time Frame: as for outcome 3
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL. Participants with no post-baseline response assessments were treated as non-responders. Four participants in the Zanubrutinib + Lenalidomide 15 mg group had a missing or unclassified GEP-subtype and are not included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- ABC Subtype: Zanubrutinib + Lenalidomide 15 mg: Participants with GEP ABC subtype received zanubrutinib 160 mg orally BID and lenalidomide 15 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- GCB Subtype: Zanubrutinib + Lenalidomide 15 mg: Participants with GEP GCB subtype received zanubrutinib 160 mg orally BID and lenalidomide 15 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- ABC Subtype: Zanubrutinib + Lenalidomide 20 mg: Participants with GEP ABC subtype received zanubrutinib 160 mg orally BID and lenalidomide 20 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- GCB Subtype: Zanubrutinib + Lenalidomide 20 mg: Participants with GEP GCB subtype received zanubrutinib 160 mg orally BID and lenalidomide 20 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- ABC Subtype: Zanubrutinib + Lenalidomide 25 mg: Participants in Part 1 with GEP ABC subtype received zanubrutinib 160 mg orally BID and lenalidomide 25 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- GCB Subtype: Zanubrutinib + Lenalidomide 25 mg: Participants in Part 1 with GEP GCB subtype received zanubrutinib 160 mg orally BID and lenalidomide 25 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
Arm/Group | ABC Subtype: Zanubrutinib + Lenalidomide 15 mg | GCB Subtype: Zanubrutinib + Lenalidomide 15 mg | ABC Subtype: Zanubrutinib + Lenalidomide 20 mg | GCB Subtype: Zanubrutinib + Lenalidomide 20 mg | ABC Subtype: Zanubrutinib + Lenalidomide 25 mg | GCB Subtype: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 1 | 1 | 8 | 2 | 9 | 2
percentage of participants | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 97.5] | 12.5 [0.3 to 52.7] | 100.0 [15.8 to 100.0] | 88.9 [51.8 to 99.7] | 100.0 [15.8 to 100.0]

28. Secondary Outcome: Part 2: Overall Response Rate by Immunohistochemistry Subtypes
Description: ORR is defined as the percentage of participants who achieved a best overall response of PR or CR based on the Lugano classification as assessed by the investigator.
  CR: complete metabolic (no/minimal FDG uptake and no evidence of FDG-avid disease in bone marrow) and radiologic response (target lesions regressed to ≤ 1.5 cm in longest diameter with no extra-lymphatic sites of disease, no organ enlargement and normal bone marrow morphology), no new lesions, and no bone marrow involvement confirmed by bone marrow biopsy (if bone marrow was involved at baseline).
  PR: partial metabolic (reduced FDG uptake from Baseline) and radiologic response (≥ 50% decrease in size of measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by > 50% in length beyond normal) and no new lesions.
  Immunohistochemistry was used to identify GCB and non-GCB phenotypes.
Time Frame: Response was assessed every 12 weeks for the first 48 weeks and every 16 weeks for the next 48 weeks and every 24 weeks thereafter; maximum time on follow-up was 31 months in the RP2D group.
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL. Participants with no post-baseline response assessments were treated as non-responders.
  For Part 2 clinical outcomes analyzed by subtype, results include all participants who received the RP2D of lenalidomide (25 mg) with non-missing subtype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- GCB Subtype: Zanubrutinib + Lenalidomide 25 mg: Participants with IHC GCB subtype who received zanubrutinib 160 mg orally BID and lenalidomide 25 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- Non-GCB Subtype: Zanubrutinib + Lenalidomide 25 mg: Participants with IHC non-GCB subtype who received zanubrutinib 160 mg orally BID and lenalidomide 25 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
Arm/Group | GCB Subtype: Zanubrutinib + Lenalidomide 25 mg | Non-GCB Subtype: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 16 | 34
percentage of participants | 50.0 [24.7 to 75.3] | 61.8 [43.6 to 77.8]

29. Secondary Outcome: Part 2: Overall Response Rate by Gene Expression Profiling Subtypes
Description: ORR is defined as the percentage of participants who achieved a best overall response of PR or CR based on the Lugano classification assessed by the investigator.
  CR: complete metabolic (no/minimal FDG uptake and no evidence of FDG-avid disease in bone marrow) and radiologic response (target lesions regressed to ≤1.5 cm in longest diameter with no extra-lymphatic sites of disease, no organ enlargement and normal bone marrow morphology), no new lesions, and no bone marrow involvement confirmed by bone marrow biopsy (if bone marrow was involved at baseline).
  PR: partial metabolic (reduced FDG uptake from Baseline) and radiologic response (≥ 50% decrease in size of measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by > 50% in length beyond normal) and no new lesions.
  Gene expression profiling by HTG EdgeSeq DLBCL COO assay was used to determine ABC and GCB subtypes.
Time Frame: as for outcome 28
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL. Participants with no post-baseline response assessments were treated as non-responders.
  For Part 2 clinical outcomes analyzed by subtype, results include all participants who received the RP2D of lenalidomide (25 mg) with non-missing subtype (four participants had a missing GEP-subtype and are not included).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- ABC Subtype: Zanubrutinib + Lenalidomide 25 mg: Participants with GEP ABC subtype who received zanubrutinib 160 mg orally BID and lenalidomide 25 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
- GCB Subtype: Zanubrutinib + Lenalidomide 25 mg: Participants with GEP GCB subtype who received zanubrutinib 160 mg orally BID and lenalidomide 25 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
Arm/Group | ABC Subtype: Zanubrutinib + Lenalidomide 25 mg | GCB Subtype: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 35 | 11
percentage of participants | 68.6 [50.7 to 83.1] | 45.5 [16.7 to 76.6]

30. Secondary Outcome: Part 2: Complete Response Rate (CRR)
Description: CRR is defined as the percentage of participants who achieved a best overall response of complete response (CR) based on the Lugano classification as assessed by the investigator. Response was evaluated using CT and metabolic imaging (FDG-PET).
  CR: complete metabolic (no/minimal FDG uptake and no evidence of FDG-avid disease in bone marrow) and radiologic response (target lesions regressed to ≤1.5 cm in longest diameter with no extra-lymphatic sites of disease, no organ enlargement and normal bone marrow morphology), no new lesions, and no bone marrow involvement confirmed by bone marrow biopsies (if bone marrow was involved at baseline).
Time Frame: as for outcome 2
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL. Participants with no post-baseline response assessments were treated as non-responders.
  Complete response rate was a prespecified secondary endpoint in Part 2 only; results are also presented for all participants who received the RP2D of lenalidomide (25 mg).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 1+2: Zanubrutinib + Lenalidomide 25 mg: All participants who received the RP2D of zanubrutinib 160 mg orally BID and lenalidomide 25 mg orally QD on Days 1-21 of each 28-day cycle until disease progression or unacceptable toxicity.
Arm/Group | Part 2: Zanubrutinib + Lenalidomide 25 mg | Part 1+2: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 39 | 50
percentage of participants | 33.3 [19.1 to 50.2] | 42.0 [28.2 to 56.8]

31. Secondary Outcome: Part 2: Complete Response Rate by Immunohistochemistry Subtypes
Description: CRR is defined as the percentage of participants who achieved a best overall response of complete response (CR) based on the Lugano classification as assessed by the investigator. Response was evaluated using CT and metabolic imaging (FDG-PET).
  CR: complete metabolic (no/minimal FDG uptake and no evidence of FDG-avid disease in bone marrow) and radiologic response (target lesions regressed to ≤1.5 cm in longest diameter with no extra-lymphatic sites of disease, no organ enlargement and normal bone marrow morphology), no new lesions, and no bone marrow involvement confirmed by bone marrow biopsies (if bone marrow was involved at baseline).
  Immunohistochemistry was used to identify GCB and non-GCB phenotypes.
Time Frame: as for outcome 28
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL. Participants with no post-baseline response assessments were treated as non-responders.
  CRR by IHC subtype was a prespecified secondary endpoint in Part 2 only. For Part 2 clinical outcomes analyzed by subtype, results include all participants who received the RP2D of lenalidomide (25 mg) with non-missing subtype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GCB Subtype: Zanubrutinib + Lenalidomide 25 mg | Non-GCB Subtype: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 16 | 34
percentage of participants | 50.0 [24.7 to 75.3] | 38.2 [22.2 to 56.4]

32. Secondary Outcome: Part 2: Complete Response Rate by Gene Expression Profiling Subtypes
Description: CRR is defined as the percentage of participants who achieved a best overall response of complete response (CR) based on the Lugano classification as assessed by the investigator. Response was evaluated using CT and metabolic imaging (FDG-PET).
  CR: complete metabolic (no/minimal FDG uptake and no evidence of FDG-avid disease in bone marrow) and radiologic response (target lesions regressed to ≤1.5 cm in longest diameter with no extra-lymphatic sites of disease, no organ enlargement and normal bone marrow morphology), no new lesions, and no bone marrow involvement confirmed by bone marrow biopsies (if bone marrow was involved at baseline).
  Gene expression profiling by HTG EdgeSeq DLBCL cell-of-origin assay was used to determine ABC and GCB subtypes.
Time Frame: as for outcome 28
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL. Participants with no post-baseline response assessments were treated as non-responders.
  CRR by GEP subtype was a prespecified secondary endpoint in Part 2 only. For Part 2 clinical outcomes analyzed by subtype, results include all participants who received the RP2D of lenalidomide (25 mg) with non-missing subtype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABC Subtype: Zanubrutinib + Lenalidomide 25 mg | GCB Subtype: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 35 | 11
percentage of participants | 45.7 [28.8 to 63.4] | 45.5 [16.7 to 76.6]

33. Secondary Outcome: Part 2: Duration of Response (DOR)
Description: DOR is defined as the time from the date that the response criteria were first met to the date that progressive disease (PD) was objectively documented or death, whichever occurred first. Median DOR was estimated using the Kaplan-Meier method. Participants who did not have disease progression were censored at their last valid assessment.
  PD: Progressive metabolic disease (increased FDG uptake from Baseline and/or new FDG-avid foci consistent with lymphoma), abnormal node or lesions with longest diameter > 1.5 cm, an increase of ≥ 50% in the product of the perpendicular diameters, and an increase in the longest diameter of 0.5 cm for lesions ≤ 2 cm or 1.0 cm for lesions > 2 cm, or any new lesions.
Time Frame: From first dose to the end of study; maximum time on follow-up was 24 months in Part 2 and 31 months in the RP2D group.
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL.
  DOR was a prespecified secondary endpoint in Part 2 only; results are also presented for all participants who received the RP2D of lenalidomide (25 mg). Participants with an overall response are included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Zanubrutinib + Lenalidomide 25 mg | Part 1+2: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 19 | 29
months | 9.10 [2.79 to NA] — "NA" indicates values that could not be estimated due to insufficient number of participants with events | 14.92 [5.45 to NA] — "NA" indicates values that could not be estimated due to insufficient number of participants with events

34. Secondary Outcome: Part 2: Duration of Response by Immunohistochemistry Subtypes
Description: DOR is defined as the time from the date that the response criteria were first met to the date that progressive disease PD was objectively documented or death, whichever occurred first. Median DOR was estimated using the Kaplan-Meier method. Participants who did not have disease progression were censored at their last valid assessment.
  Immunohistochemistry was used to identify GCB and non-GCB phenotypes.
Time Frame: From first dose to the end of study; maximum time on follow-up was 31 months in the RP2D group.
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL.
  DOR by IHC subtype was a prespecified secondary endpoint in Part 2 only. For Part 2 clinical outcomes analyzed by subtype, results include all participants who received the RP2D of lenalidomide (25 mg). Participants with an overall response and non-missing IHC subtype are included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GCB Subtype: Zanubrutinib + Lenalidomide 25 mg | Non-GCB Subtype: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 8 | 21
months | NA [2.76 to NA] — "NA" indicates values that could not be estimated due to insufficient number of participants with events | 11.61 [2.83 to NA] — "NA" indicates values that could not be estimated due to insufficient number of participants with events

35. Secondary Outcome: Part 2: Duration of Response by Gene Expression Profiling Subtypes
Description: DOR is defined as the time from the date that the response criteria were first met to the date that progressive disease PD was objectively documented or death, whichever occurred first. Median DOR was estimated using the Kaplan-Meier method. Participants who did not have disease progression were censored at their last valid assessment.
  Gene expression profiling by HTG EdgeSeq DLBCL cell-of-origin assay was used to determine ABC and GCB subtypes.
Time Frame: From first dose to the end of study; maximum time on follow-up was 31 months in the RP2D group.
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL.
  DOR by GEP subtype was a prespecified secondary endpoint in Part 2 only. For Part 2 clinical outcomes analyzed by subtype, results include all participants who received the RP2D of lenalidomide (25 mg). Participants with an overall response and non-missing GEP subtype are included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABC Subtype: Zanubrutinib + Lenalidomide 25 mg | GCB Subtype: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 24 | 5
months | 15.67 [3.02 to NA] — "NA" indicates values that could not be estimated due to insufficient number of participants with events | 9.10 [3.02 to NA] — "NA" indicates values that could not be estimated due to insufficient number of participants with events

36. Secondary Outcome: Part 2: Progression-free Survival (PFS)
Description: PFS is defined as the time from the starting date of the combination therapy to the date of first documentation of disease progression or death, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Participants who did not have disease progression were censored at their last valid tumor assessment.
Time Frame: From first dose to the end of study; maximum time on follow-up was 24 months in Part 2 and 31 months in the RP2D group.
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL.
  PFS was a prespecified secondary endpoint in Part 2 only; results are also presented for all participants who received the RP2D of lenalidomide.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: Zanubrutinib + Lenalidomide 25 mg | Part 1+2: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 39 | 50
months | 4.76 [2.73 to 8.94] | 5.52 [2.86 to 11.07]

37. Secondary Outcome: Part 2: Progression-Free Survival by Immunohistochemistry Subtypes
Description: PFS is defined as the time from the starting date of the combination therapy to the date of first documentation of disease progression or death, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Participants who did not have disease progression were censored at their last valid tumor assessment.
  Immunohistochemistry was used to identify GCB and non-GCB phenotypes.
Time Frame: From first dose to the end of study; maximum time on follow-up was 31 months in the RP2D group.
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL.
  PFS by IHC subtype was a prespecified secondary endpoint in Part 2 only. For Part 2 clinical outcomes analyzed by subtype, results include all participants who received the RP2D of lenalidomide (25 mg) with non-missing subtype.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GCB Subtype: Zanubrutinib + Lenalidomide 25 mg | Non-GCB Subtype: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 16 | 34
months | 5.55 [1.61 to NA] — "NA" indicates values that could not be estimated due to insufficient number of participants with events | 5.52 [2.86 to 11.04]

38. Secondary Outcome: Part 2: Progression-Free Survival by Gene Expression Profiling Subtypes
Description: PFS is defined as the time from the starting date of the combination therapy to the date of first documentation of disease progression or death, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Participants who did not have disease progression were censored at their last valid tumor assessment.
  Gene expression profiling by HTG EdgeSeq DLBCL cell-of-origin assay was used to determine ABC and GCB subtypes.
Time Frame: From first dose to the end of study; maximum time on follow-up was 31 months in the RP2D group.
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL.
  PFS by GEP subtype was a prespecified secondary endpoint in Part 2 only. For Part 2 clinical outcomes analyzed by subtype, results include all participants who received the RP2D of lenalidomide (25 mg) with non-missing subtype (four participants had a missing GEP-subtype and are not included).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABC Subtype: Zanubrutinib + Lenalidomide 25 mg | GCB Subtype: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 35 | 11
months | 5.55 [4.76 to 18.40] | 5.40 [1.41 to 14.65]

39. Secondary Outcome: Part 2: Time to Response (TTR)
Description: Time to response is defined as time from the starting date of combination therapy to the date the response criteria were first met.
Time Frame: as for outcome 2
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL.
  TTR was a prespecified secondary endpoint in Part 2 only; results are also presented for all participants who received the RP2D of lenalidomide (25 mg). Participants with an overall response are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Part 2: Zanubrutinib + Lenalidomide 25 mg | Part 1+2: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 19 | 29
months | 2.76 [2.73 to 2.89] | 2.76 [2.73 to 2.83]

40. Secondary Outcome: Part 2: Time to Response by Immunohistochemistry Subtypes
Description: Time to response is defined as time from the starting date of combination therapy to the date the response criteria were first met.
  Immunohistochemistry was used to identify GCB and non-GCB phenotypes.
Time Frame: as for outcome 28
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL.
  TTR by IHC subtype was a prespecified secondary endpoint in Part 2 only. For Part 2 clinical outcomes analyzed by subtype, results include all participants who received the RP2D of lenalidomide (25 mg). Participants with an overall response and non-missing IHC subtype are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | GCB Subtype: Zanubrutinib + Lenalidomide 25 mg | Non-GCB Subtype: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 8 | 21
months | 2.87 [2.78 to 3.33] | 2.76 [2.73 to 2.79]

41. Secondary Outcome: Part 2: Time to Response by Gene Expression Profiling Subtypes
Description: Time to response is defined as the time from the starting date of combination therapy to the date objective response criteria were first met.
  Gene expression profiling by HTG EdgeSeq DLBCL cell-of-origin assay was used to determine ABC and GCB subtypes.
Time Frame: From first dose to the end of study; maximum time on follow-up was 31 months in the RP2D group.
Population: The efficacy analysis set was defined as all participants who were exposed to at least one dose of medication with confirmed R/R DLBCL.
  TTR by GEP subtype was a prespecified secondary endpoint in Part 2 only. For Part 2 clinical outcomes analyzed by subtype, results include all participants who received the RP2D of lenalidomide (25 mg). Participants with an overall response and non-missing GEP subtype are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | ABC Subtype: Zanubrutinib + Lenalidomide 25 mg | GCB Subtype: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 24 | 5
months | 2.76 [2.73 to 2.83] | 3.19 [2.79 to 3.48]

42. Secondary Outcome: Part 2: Number of Participants With Treatment-emergent Adverse Events
Description: An AE is defined as any untoward medical occurrence in a patient temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product (zanubrutinib in combination with lenalidomide).
  A serious adverse event (SAE) is any untoward medical occurrence that, at any dose:
  * Resulted in death.
  * Was life threatening.
  * Required hospitalization or prolongation of existing hospitalization.
  * Resulted in disability/incapacity.
  * Was a congenital anomaly/birth defect.
  * Was considered a significant medical AE by the investigator based on medical judgement (eg, may have jeopardized the patient or may have required medical/surgical intervention to prevent one of the outcomes listed above).
Time Frame: From first dose of study drug to 30 days after last dose. Maximum time on treatment in Part 2 was 701 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Zanubrutinib + Lenalidomide 25 mg
Number analyzed (Participants) | 39
Participants
  TEAEs | 39
  SAEs | 14

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to the end of study, maximum time on study was 41.6 months. AEs: From first dose of study drug to 30 days after last dose. Maximum time on treatment was 1260 days.
Arm/Group | Part 1: Zanubrutinib + Lenalidomide 15 mg | Part 1: Zanubrutinib + Lenalidomide 20 mg | Part 1: Zanubrutinib + Lenalidomide 25 mg | Part 2: Zanubrutinib + Lenalidomide 25 mg
All-Cause Mortality (participants affected / at risk) | 3/6 | 5/10 | 3/11 | 18/39
Serious Adverse Events (participants affected / at risk) | 0/6 | 3/10 | 4/11 | 14/39
Other Adverse Events (participants affected / at risk) | 6/6 | 10/10 | 11/11 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Zanubrutinib + Lenalidomide 15 mg (N=6) | Part 1: Zanubrutinib + Lenalidomide 20 mg (N=10) | Part 1: Zanubrutinib + Lenalidomide 25 mg (N=11) | Part 2: Zanubrutinib + Lenalidomide 25 mg (N=39)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pneumonia (Infections and infestations) | 0 (0) | 2 (3) | 2 (8) | 4 (9)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 1 (3) | 2 (4)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (26) | 2 (12)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scalp haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Zanubrutinib + Lenalidomide 15 mg (N=6) | Part 1: Zanubrutinib + Lenalidomide 20 mg (N=10) | Part 1: Zanubrutinib + Lenalidomide 25 mg (N=11) | Part 2: Zanubrutinib + Lenalidomide 25 mg (N=39)
Anaemia (Blood and lymphatic system disorders) | 2 (9) | 4 (20) | 8 (43) | 21 (65)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (7) | 0 (0) | 1 (1) | 2 (5)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (9) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (6) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Thyroid cyst (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 2 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (4) | 1 (2) | 0 (0) | 4 (6)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (2) | 1 (1) | 5 (6)
Asthenia (General disorders) | 2 (2) | 1 (1) | 1 (1) | 5 (7)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (5) | 3 (5)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (8)
Peripheral swelling (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (4) | 3 (5) | 5 (6)
Swelling face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 9 (11)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cervicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (7) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (4) | 5 (7) | 10 (21)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (4) | 5 (7) | 9 (19)
Basophil count increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Beta 2 microglobulin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 6 (10)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 2 (5) | 2 (2) | 9 (11)
Blood bilirubin increased (Investigations) | 1 (3) | 0 (0) | 2 (4) | 9 (23)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 2 (4)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 3 (3) | 1 (2) | 9 (19)
Blood fibrinogen decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood fibrinogen increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 2 (4) | 6 (7) | 1 (1) | 13 (14)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 8 (12)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eosinophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 2 (3) | 2 (2) | 5 (7)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (2) | 4 (8) | 11 (15)
Globulins decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 4 (25) | 5 (28) | 6 (64) | 14 (50)
Monocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (29) | 6 (44) | 10 (117) | 33 (283)
Platelet count decreased (Investigations) | 2 (2) | 7 (39) | 6 (64) | 24 (105)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 3 (5) | 2 (3) | 1 (1) | 3 (4)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
White blood cell count decreased (Investigations) | 3 (18) | 6 (33) | 10 (117) | 29 (176)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (6)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0) | 4 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (6) | 8 (14)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (5) | 1 (1) | 4 (9)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (7) | 0 (0) | 6 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (8) | 3 (10) | 11 (21)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 3 (4) | 7 (12)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 4 (6) | 6 (23) | 15 (35)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 2 (4) | 3 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 2 (2) | 7 (11)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (9) | 1 (3)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 1 (2) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (4)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epididymal cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Cystic lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 2 (2) | 12 (20)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (6)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (6) | 3 (7)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period,Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT04436107/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT04436107/SAP_001.pdf